CLINICAL TRIAL: NCT02306525
Title: Outcome After Arthroscopic Treatment of Patients in Horsens and Aarhus With FemoroAcetabular Impingement: the HAFAI-cohort
Brief Title: Arthroscopic Treatment of Patients in Horsens and Aarhus With FemoroAcetabular Impingement: the HAFAI-cohort
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Horsens Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-239-14; 1-16-02-499-14 (Other: The Danish Data Protection Agency)
Record Dates: First submitted 2014-11-21; First posted 2014-12-03 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Femoracetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Ptt. with Femoracetabular Impingement: Enrollment anticipated: 60 Arthroscopic surgery of the hip joint
  Interventions: Procedure: Arthroscopic surgery of the hip joint
- Healthy volunteers: Enrollment anticipated: 30

INTERVENTIONS:
Procedure: Arthroscopic surgery of the hip joint — Arthroscopic treatment of Femoroacetabular Impingement
  Other Names: Hip Arthroscopy; Arthroscopic surgery of Femoro-Acetabular Impingement
  Groups: Ptt. with Femoracetabular Impingement

SUMMARY:
Purpose: The aim of this prospective cohort is to evaluate patients before, 6 and 12 months after arthroscopic surgery for FAI and compare the results to people without hip problems.

Methods/design: Sixty patients with FAI and 30 persons without hip problems will be included. Pre- and postoperatively, patients will be evaluated by CT-scans. All participants will have their hip flexor and extensor muscle strength assessed and have performed kinetic and kinematic analyses of daily activities with 3D motion capture. Further, self-reported questionnaires on hip related pain, quality of life and sports activities will be collected. Finally, participants will have their daily physical activity monitored with tri-axial accelerometers for five consecutive days.

Perspectives: With this prospective cohort study the outcome of arthroscopic treatment of FAI within one year after surgery will be evaluated. If the patients fail to reach reference values one year after surgery, altered surgical procedures or rehabilitation programs to optimize treatment for the patients may be explored in future studies. Further, the investigators expect to perform long-term follow up to evaluate reoperations, conversions to total hip arthroplasty and development of osteoarthritis for the patients surgically treated for FAI.

DETAILED DESCRIPTION:
Introduction Femoral acetabular impingement (FAI) is caused by an abnormality in the acetabular shape or orientation (Pincer-type) by a shape abnormality in the proximal femur (Cam-type) or by a mix of the two conditions. FAI causes repeated minor damage to the labrum and edge of the acetabulum. The damage to the joint is proposed to lead to early osteoarthritis (OA) of the hip, but whether FAI is a cause or result of OA is discussed. Surgery can reduce symptoms caused by Cam or Pincer impingement and may prevent future damage to the hip joint. However, different surgical techniques are used, and only few long-term studies of the surgery exist. The latest reviews conclude that 1) the effectiveness of the surgery is not clear, 2) it is not clear how surgery affects functional performance for the patients and 3) it is unknown how surgery for FAI affects the patients in a long-term perspective.

Material and methods

Patients:

Inclusion criteria

* Planned hip arthroscopic treatment at Horsens Regional Hospital by Consultant Bent Lund
* A diagnosis of CAM and/or pincer impingement
* For patients with Cam, an alpha angle > 55 degrees on an anterior/posterior (AP) standing radiograph
* For patients with Pincer a center edge angle > 25 degrees on an AP radiograph
* No signs of retroversion in the lower 2/3 of the hip joint on an AP radiograph
* No posterior wall sign on an AP radiograph
* Osteoarthritis grade 0-1 according to Tönnis' classification
* Lateral Joint space width of > 3 mm
* Age between 18 and 50 years

Exclusion criteria

* Previous hip operations of the included hip
* Persons with FAI secondary to other hip conditions such as Calvé Perthes and epiphysiolysis.
* Alloplastic surgery at the hip, knee or ankle region (both legs)
* Neurological diseases
* Cancer
* Inability to speak or understand Danish
* Pregnancy at the time of inclusion

Control persons (healthy volunteers) Thirty gender and age-matched persons with no known hip, knee or ankle region problems will be included as controls.

Primary outcome measures

* Hip and pelvis kinetics and kinematics during walking, stair climbing, stepping, sit-to-stand and drop jump
* Hip extensor and flexor maximal muscle strength during isometric and isokinetic contractions
* Hip extensor and flexor rate of force development during isometric contraction
* Objectively measured daily physical activities during 5 days
* Hip- related self-reported health measured with the Copenhagen Hip and Groin Outcome Score

Secondary outcome measures

* Knee and trunk kinetics and kinematics during walking, stair climbing, stepping, sit-to-stand and jump
* Hip extensor and flexor rate of force development during isometric contraction
* Self-selected walking speed
* Presence of intra-articular pathology examined with FABER and impingement tests
* Visual analog scale, pain
* Patient expectations
* Reasons for choosing surgery
* Patient global treatment outcome
* Patient-acceptable symptom state
* EQ5D-Visual analog scale
* Failure
* Re-operations and injections during the first year after surgery
* Self-reported present sports activities
* Time spend at preferred sports activity present
* Time spend at sports activities during childhood
* Sports activities during childhood
* Return to sports activities
* Education
* Employment
* Smoking habits
* Alcohol intake
* Intake of analgesia
* Comorbidities

Other Pre-specified Outcome Measures:

* Alpha angle
* Wiberg's center-edge (CE) angle
* Tönnis' acetabular index (AI)
* Retroversion of acetabulum
* The position of the femoral head in relation to the neck
* Osteoarthritis grade according to Tönnis' classification
* Lateral hip joint space width
* Information about the surgical procedure immediately
* Deviation from rehabilitation program
* Duration of pain
* Body Mass Index
* Body fat percentage
* Age

Procedure

Patients scheduled for hip arthroscopic treatment at Horsens Regional Hospital will receive written and verbal information about the study and after informed consent included consecutively. After agreeing to participate, the patients will have a pre-operative CT-scan of the included hip. At Aarhus University, patients will have a clinical examination session including measurement of height, weight and fat percentage. They will have their hip extensor and flexor muscle strength assessed in an isokinetic dynamometer and perform walking, stair climbing, stepping, sit to stand and a drop jump with 3D-motion capture. Patients will complete the HAGOS-questionnaire together with the other pre specified self-reported measures described.

After all tests are completed, the patients will be instructed in wearing a 3-axial accelerometer for five days, attached to the thigh of the non-affected leg to monitor daily physical activity.

At a three, six and nine month follow-up patients will complete HAGOS, pain scores and self-reported measures of return to sport, work, re-operations and injections after surgery and EQ5D-Visual analog scale.

At a one year follow up, preoperative measures will be repeated. Further, at six month and one year follow up the patients will report fulfillment of expectations, patient global treatment outcome and patient willingness to repeat surgery.

All controls will meet at Aarhus University for a single assessment of the same measures as the patients except from CT-scans and outcome measures related to the surgery.

Statistics

Patients and controls will be compared with multiple regression analysis adjusted for age, gender and body weight if the assumptions for the model is met. If not, they will be compared using un-paired non-parametric statistics.

The longitudinal measures of the patients pre, three, six, nine month and one year after surgery will be evaluated in a paired set-up.

Further analyses

Based upon the preoperative CT-scan, the patients will be split into subgroups: FAI will be classified as Cam (alpha angle > 55˚), Pincer (center edge angle > 25˚ from CT and AP radiograph and/or crossing sign and ishial spine sign) and Mixed when there is a combination of Cam and Pincer. We will investigate how these subgroups affects outcome measures. Further, we will investigate how demographics, preoperative and postoperative muscle strength and pain affects the results of the surgery and rehabilitation procedure.

Sample size

The primary end point for the study is one year after surgery. For the muscle strength assessment, sample size is based upon pre- and post-operative values from Casartelli et al. (2) with a level of significance of 0.05 and a power of 90 %, the patient group should consist at least 53 persons. Taking possible drop-outs in account our goal is to include 60 patients. We will include 30 controls persons for comparisons.

Ethics

The Danish Biomedical Research Ethics Committee, Central Denmark Region (1-10-72-239-14) and the Danish Data Protection Agency have approved the project (1-16-02-499-14).

Economy and dissemination

Financial support will be applied for at internally at our institution and externally at various foundations. Both positive, negative and inconclusive results will be published in international journals and presented at conferences.

References

1. Mannion AF, Impellizzeri FM, Naal FD, Leunig M: Fulfilment of patient-rated expectations predicts the outcome of surgery for femoroacetabular impingement. Osteoarthritis and Cartilage 2013, 21:44-50.
2. Casartelli NC, Maffiuletti NA, Item-Glatthorn JF, Impellizzeri FM, Leunig M: Hip muscle strength recovery after hip arthroscopy in a series of patients with symptomatic femoroacetabular impingement. Hip international : the journal of clinical and experimental research on hip pathology and therapy 2014:0.
3. Paulsen A, Roos EM, Pedersen AB, Overgaard S. Minimal clinically important improvement (MCII) and patient-acceptable symptom state (PASS) in total hip arthroplasty (THA) patients 1 year postoperatively. Acta orthopaedica. 2014;85(1):39-48.

ELIGIBILITY:
Inclusion Criteria (patients):

* Planned hip arthroscopic treatment at Horsens Regional Hospital by Consultant Bent Lund
* A diagnosis of CAM and/or pincer impingement
* For patients with Cam, an alpha angle > 55 degrees on an anterior/posterior (AP) standing radiograph
* For patients with Pincer a center edge angle > 25 degrees on an AP radiograph
* No signs of retroversion in the lower 2/3 of the hip joint on an AP radiograph
* No posterior wall sign on an AP radiograph
* Osteoarthritis grade 0-1 according to Tönnis' classification
* Lateral Joint space width of > 3 mm
* Age between 18 and 50 years

Exclusion Criteria (patients):

* Previous hip operations of the included hip
* Persons with FAI secondary to other hip conditions such as Calvé Perthes and epiphysiolysis.
* Alloplastic surgery at the hip, knee or ankle region (both legs)
* Neurological diseases
* Cancer
* Inability to speak or understand Danish
* Pregnancy at the time of inclusion

Control persons (healthy volunteers):

* Gender and age-matched persons
* No known hip, knee or ankle region problems

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with Femoro Acetabular Impingement and Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Hip and pelvis kinetics and kinematics during walking, stair climbing, stepping, sit-to-stand and drop jump | Change from preoperatively (Approx. in the time frame 0-10 weeks before surgery) to one year after surgery
  Hip and pelvis kinetics and kinematics are measured with a 3D motion capture system with a force platform using a standardized protocol
Hip extensor and flexor maximal muscle strength during isometric and isokinetic contractions | Change from preoperatively (Approx. in the time frame 0-10 weeks before surgery) to one year after surgery
  Hip extensor and flexor maximal strength is measured with an isokinetic dynamometer using a standardized protocol
Objectively measured daily physical activities during five days | Change from preoperatively (Approx. in the time frame 0-10 weeks before surgery) to one year after surgery
  Physical activity is measured with a tri-axial accelerometer during a period of 5 days on the following categories: rest, standing, walking, sit to stand, cycling and high impact activity.
Hip-related self-reported health | Change from preoperatively (Approx. in the time frame 0-10 weeks before surgery) to one year after surgery
  Hip related health is measured with the Copenhagen Hip and Groin Outcome Score (HAGOS) validated on patients with hip and groin pain

SECONDARY OUTCOMES:
Knee and trunk kinetics and kinematics during walking, stair climbing, stepping, sit-to-stand drop jump | Preoperatively (Approx. in the time frame 0-10 weeks before surgery) and one year after surgery
  Knee and trunk kinetics and kinematics are measured with a 3D motion capture system with a force platform using a standardized protocol
Hip extensor and flexor rate of force development during isometric contraction | Preoperatively (Approx. in the time frame 0-10 weeks before surgery) and one year after surgery
  Hip extensor and flexor rate of force development is measured with an isokinetic dynamometer using a standardized protocol
Self-selected walking speed | Preoperatively (Approx. in the time frame 0-10 weeks before surgery) and one year after surgery
Presence of intra-articular pathology examined with FABER and impingement tests | Preoperatively (Approx. in the time frame 0-10 weeks before surgery) and one year after surgery
Visual analog scale, pain | Preoperatively (Approx. in the time frame 0-10 weeks before surgery) and one year after surgery
  Pain is measured during rest and activity with a visual analog scale. Further patients will report their pain at a visual analog scale during all physical performance tests
Patient expectations | Preoperatively (Approx. in the time frame 0-10 weeks before surgery), 6 month and one year after surgery
  The question, "what changes in the following items do you expect to experience as a result of the operation? (not your hopes and wishes, but realistic expectations!)" will be asked in relation to each of six items: hip pain, walking capacity, independence in everyday activities, ability to do sport, engaging in social contacts, mental well-being. The response options will be: much better, better, somewhat better, unchanged, worse, "I don't know". After surgery, the same response options will be given together with the question: "what changes in the following items have occurred as a result of the operation?" (Adapted from Mannion et al. (1))
Reasons for choosing surgery | Preoperatively (Approx. in the time frame 0-10 weeks before surgery)
Patient global treatment outcome | Six month and one year after surgery
  The question: "How much did the operation help your hip problem?" will be asked together with the options: helped a lot, helped, helped only little, didn't help, made things worse. Adapted from Mannion et al. (1)
Patient-acceptable symptom state | Six month and one year after surgery
  The question "How would you describe the result of your operation?" will be asked. There will be 5 response options: "Excellent", "Very good", "Good", "Fair", and "Poor". Adapted from Paulsen et al. (3)
EQ5D-Visual analog scale | Preoperatively (Approx. in the time frame 0-10 weeks before surgery), 6 month and one year after surgery
  Overall health will be evaluated with the EQ5D- Visual analog scale
Failure | One year after surgery
  The surgical treatment and rehabilitation will be considered a failure if the patient have received a total hip arthroplasty
Re-operations and injections during the first year after surgery | 3 month, 6 month, 9 month and one year after surgery
Self-reported present sports activities | Preoperatively (Approx. in the time frame 0-10 weeks before surgery), 3 month, 6 month, 9 month and one year after surgery
Time spend at preferred sports activity | Preoperatively (Approx. in the time frame 0-10 weeks before surgery), 3 month, 6 month, 9 month and one year after surgery
Sports activities during childhood (age < 18) | Preoperatively (Approx. in the time frame 0-10 weeks before surgery)
Time spend at sports activities during childhood | Preoperatively (Approx. in the time frame 0-10 weeks before surgery)
Education | Preoperatively (Approx. i the time frame 0-10 weeks before surgery)
Employment | Preoperatively (Approx. in the time frame 0-10 weeks before surgery)
Smoking habits | Preoperatively (Approx. in the time frame 0-10 weeks before surgery), one year after surgery
Alcohol intake | Preoperatively (Approx. in the time frame 0-10 weeks before surgery), one year after surgery
Intake of analgesia | Preoperatively (Approx. in the time frame 0-10 weeks before surgery), 3 month, 6 month, 9 month and one year after surgery
Comorbidities | Preoperatively (Approx. in the time frame 0-10 weeks before surgery)
  Patients will report comorbidities as hypertension, diabetes ect.

OTHER OUTCOMES:
Alpha angle | Preoperatively (Approx. in the time frame 0-10 weeks before surgery) and one year after surgery
Wiberg's center-edge (CE) angle | Prior to surgery (Preoperatively (Approx. in the time frame 0-10 weeks before surgery)and one year after surgery
Tönnis' acetabular index (AI) | Preoperatively (Approx. in the time frame 0-10 weeks before surgery) and one year after surgery
Retroversion of acetabulum | Preoperatively (Approx. in the time frame 0-10 weeks before surgery) and one year after surgery
  Measured at low dosis CT-scans
The position of the femoral head in relation to the neck | Preoperatively (Approx. in the time frame 0-10 weeks before surgery) and one year after surgery
  Measured at low dosis CT-scans
Osteoarthritis grade according to Tönnis' classification | Preoperatively (Approx. in the time frame 0-10 weeks before surgery) and one year after surgery
Lateral hip joint space width | Preoperatively (Approx. in the time frame 0-10 weeks before surgery) and one year after surgery
Information about the surgical procedure | Immediately after completing surgical procedure
  Described by the surgeon after leaving the operation theater
Deviation from rehabilitation program | During the rehabilitation period that lasts around 1 year
  Deviation from rehabilitation program will be recorded by physiotherapists
Duration of pain | Preoperatively (Approx. in the time frame 0-10 weeks before surgery)
Body Mass Index | Preoperatively (Approx. in the time frame 0-10 weeks before surgery) and one year after surgery
Body fat percentage | Preoperatively (Approx. in the time frame 0-10 weeks before surgery) and one year after surgery
Age | Preoperatively (Approx. in the time frame 0-10 weeks before surgery)
Hip-related self-reported health | 3, 6 and 9 months after surgery
  Hip related health is measured with the Copenhagen Hip and Groin Outcome Score (HAGOS) validated on patients with hip and groin pain

CONTACTS AND LOCATIONS:
Overall Officials: Inger Mechlenburg, PhD, Study Director — Orthopedic Research, Aarhus University and University Hospital, Denmark; Kjeld Søballe, Professor,MD, Study Chair — Orthopedic Research, Aarhus University and University Hospital, Denmark; Ulrik Dalgas, PhD, Study Chair — Section of Sport, Aarhus University, Denmark; Bent Lund, MD, Study Chair — Horsens Regional Hospital, Denmark; Henrik Sørensen, PhD, Study Chair — Section of Sport, Aarhus University, Denmark; Lone Rømer, MD, Study Chair — Aarhus University Hospital, Denmark
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus, DK
  - Section of Sport, Aarhus University, Aarhus, DK
  - Horsens Regional Hospital, Horsens, DK

REFERENCES:
- [Derived] Kierkegaard S, Lund B, Dalgas U, Sorensen H, Soballe K, Mechlenburg I. The Horsens-Aarhus Femoro Acetabular Impingement (HAFAI) cohort: outcome of arthroscopic treatment for femoroacetabular impingement. Protocol for a prospective cohort study. BMJ Open. 2015 Sep 7;5(9):e008952. doi: 10.1136/bmjopen-2015-008952. PMID 26346877